CLINICAL TRIAL: NCT03359031
Title: Effects of Perioperative Patient Education Regarding Compartment Syndrome on Post-operative Opioid Consumption
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-Krieg
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Compartment Syndrome of Leg
MeSH Terms: interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No patient education (No Intervention): This group of patients will not receive any additional information beyond standard of care educational pamphlets provided by the hospital.
- Patient education (Other): This group of patients will be given a pamphlet on pain control, narcotic medication, and compartment syndrome including its pathophysiology, signs/symptoms, and treatment.
  Interventions: Other: Patient education

INTERVENTIONS:
Other: Patient education — This group will be given a pamphlet on pain control, narcotic medication, and compartment syndrome including its pathophysiology, signs/symptoms, and treatment.
  Arms: Patient education

SUMMARY:
This study is a prospective, randomized trial. Our study aims to study the effects of perioperative patient education about compartment syndrome on patients' perception of their own pain, amount of opioid medication utilization, and rate of diagnosis of compartment syndrome.

ELIGIBILITY:
Inclusion Criteria:

Patients with lower extremity trauma at risk for developing compartment syndrome specifically tibial plateau fractures, tibial/fibular shaft fractures, pilon fractures, and crush injuries.

Exclusion Criteria:

Patients with an extensive history of narcotic medication or drug use, polytrauma patients, and non-primary English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
narcotic consumption | total opioid consumption from surgery through 30 days post-op
  Perioperative

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No